CLINICAL TRIAL: NCT05750901
Title: Pilot Evaluation of Fractional Ablative Laser Treatment for Skin Laxity and Tightening
Brief Title: Evaluation of Fractional Ablative Laser Treatment for Skin Conditions
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sciton (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LC-001
Record Dates: First submitted 2023-02-08; First posted 2023-03-02 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Treatment Arm (Other): Patients will receive fractional ablative treatment for laxity.
  Interventions: Device: Fractional ablative laser

INTERVENTIONS:
Device: Fractional ablative laser — Fractional ablative laser used for treatment for skin laxity and tightening

SUMMARY:
Evaluate the safety and efficacy of the fractional ablative laser for treatment of skin laxity and tightening

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects aged 18-85 years
2. Fitzpatrick skin type I-VI
3. Has visible skin laxity in the treatment region or has a scar
4. Post-menopausal or surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrollment and during the entire course of the study, and no plans to become pregnant for the duration of the study (Applicable to female subjects only)
5. Willing to have digital imaging and measurements taken of the treatment area and agree to use for presentation, educational or marketing purposes
6. Subject must be able to read, understand and sign Informed Consent Form in English
7. Must be willing to adhere to the treatment and follow-up schedule and post-treatment care instructions

Exclusion Criteria:

1. Participation in a clinical trial of another device or drug within 6 months prior to enrollment or during the study.
2. Any type of prior cosmetic treatment to the target area at physicians' discretion
3. History of malignant tumors in the target area.
4. Skin abnormalities in the target area, e.g., cuts, scrapes, wounds, large moles.
5. Pregnant and/or breastfeeding (Applicable to females only)
6. Having an infection, dermatitis or a rash in the treatment area.
7. Significant concurrent illness, such as diabetes mellitus, cardiovascular disease, e.g., uncontrolled hypertension or pertinent neurological disorders.
8. Suffering from coagulation disorders or taking prescription anticoagulation medications.
9. History of keloid scarring, hypertrophic scarring or of abnormal wound healing.
10. History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications.
11. History of vitiligo, eczema, or psoriasis.
12. History of disease stimulated by heat, such as recurrent herpes simplex and/or herpes zoster (shingles) in the treatment area, unless treatment is conducted following a prophylactic regimen.
13. History of radiation to the treatment area or undergoing systemic chemotherapy for the treatment of cancer.
14. Current smoker or history of smoking within 6 months of study participation.
15. As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in this study

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-11-01 (Actual); Primary Completion 2026-03-30 (Estimated); Study Completion 2026-06-20 (Estimated)

PRIMARY OUTCOMES:
Wrinkles | 1-6 months post final treatment
  Percent improvement in wrinkles will be assessed using digital camera at baseline and post final treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Sanctuary Plastic Surgery, Boca Raton, Florida, United States